CLINICAL TRIAL: NCT02809066
Title: Effect of Sufficient Dietary Calcium Intake in Women With Premenstrual Syndrome
Brief Title: Dietary Calcium Intake in Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Merve YURT, Senior Instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/10-03
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Premenstrual Syndrome
Keywords: premenstrual syndrome; calcium; quality of life
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional group (Experimental): 8-week follow- up with dietary sufficient calcium intake
  Interventions: Other: Sufficient dietary calcium intake in premenstrual syndrome
- Control group (No Intervention): 8-week follow- up with no specific diet

INTERVENTIONS:
Other: Sufficient dietary calcium intake in premenstrual syndrome — Intervention group was ensured to take at least 1000 mg calcium from foods, 700-800 mg of it from dairy and dairy products, according to Recommended Dietary Allowances (RDA), for two months. These foods were;
  * 50 gr kashkaval cheese,
  * 400 ml milk and
  * 150 gr yogurt for each day.
  Arms: Interventional group

SUMMARY:
This study was planned and conducted to investigate effect of adequate calcium intake on Premenstrual Syndrome (PMS) symptoms in women with PMS who have inadequate calcium intake.

DETAILED DESCRIPTION:
This study was planned and conducted to investigate effect of adequate calcium intake on Premenstrual Syndrome (PMS) symptoms in women with PMS who have inadequate calcium intake. Thirty one women, aged between 20-28 years, diagnosed with PMS and suitable for inclusion criteria, were participated in study. Participants were allocated to intervention (n=16) and control (n=15) groups randomly.

ELIGIBILITY:
Inclusion Criteria:

Women with;

* PMS who have inadequate calcium intake
* Regular menstrual cycle
* Menstrual flow which occurs every 22 to 35 days and last three to eight days

Exclusion Criteria:

* Having any of metabolic diseases
* Use oral contraceptive pill
* user vitamins and minerals supplements
* being smoker

Ages: 20 Years to 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Premenstrual Syndrome Scale (PMSS) | Eight weeks
  Premenstrual Syndrome Scale (PMSS) was used for symptom assessment at initial and after two menstrual cycles.

SECONDARY OUTCOMES:
Change in Quality of life scale Short Form (SF-36) | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yurt, MS, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided